CLINICAL TRIAL: NCT06298578
Title: The Utility of Mobile Based Application for Patient Reported Outcome Measures In Patients With Acetabular Fractures : A Randomized Clinical Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Adly Attia Ayoub, Resident, Assiut University
Other Study IDs: Mobile Based Application
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In person follow up
- mobile app follow up

SUMMARY:
The primary objective of this study is to validate the feasibility of a remote patient monitoring (RPM) system using Mobile App in terms of the frequency of data interruptions and patient acceptance.

The secondary objective is to Improve quality of life and early prediction of the complications.

DETAILED DESCRIPTION:
Acetabular fractures are articular fractures involving the hip joint that needs anatomical reduction and a strict long follow up after fixation. The percentage of patients with lost follow up is significantly high. Previously all other studies mainly focused on the radiographic outcome after acetabular fractures and rarely on patient reported functional outcomes and quality of life.The use of patient-reported outcome measures (PROMs) is increasing and may lead to modifications of treatment. Recent technologic advances, namely smartphones, capable of measuring outcomes after acetabular fractures are now very important in quantifying value-based care. This was previously accomplished through office assessments and surveys with variable follow-up, but this strategy lacks continuous and complete data. Studies show that these remote modes of follow-up are safe and that patients are as equally satisfied with them as they are with in-person follow- up care.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged more than 18 years who will have a surgery for an acetabular fracture at assiut university hospital.

Exclusion Criteria:

* Patients younger than 18years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged more than 18 years who will have a surgery for an acetabular fracture at assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
percentage of missed follow up data in both groups postoperatively through assessing the patient-reported outcome measures (PROMS) after surgery for a fracture of the acetabulum using the Arabic validated form of (SF-36) | Baseline
  Comparison between follow up using mobile app versus in person clinic visit

SECONDARY OUTCOMES:
Quality of life scoring (Arabic validated form of (SF-36) and early prediction of the complications | Baseline
  Scoring postoperative quality of life and eary detection of complications

REFERENCES:
- [Background] JUDET R, JUDET J, LETOURNEL E. FRACTURES OF THE ACETABULUM: CLASSIFICATION AND SURGICAL APPROACHES FOR OPEN REDUCTION. PRELIMINARY REPORT. J Bone Joint Surg Am. 1964 Dec;46:1615-46. No abstract available. PMID 14239854
- [Background] Mears DC, Velyvis JH, Chang CP. Displaced acetabular fractures managed operatively: indicators of outcome. Clin Orthop Relat Res. 2003 Feb;(407):173-86. doi: 10.1097/00003086-200302000-00026. PMID 12567145
- [Background] Frietman B, Biert J, Edwards MJR. Patient-reported outcome measures after surgery for an acetabular fracture. Bone Joint J. 2018 May 1;100-B(5):640-645. doi: 10.1302/0301-620X.100B5.BJJ-2017-0871.R3. PMID 29701094
- [Background] Giannoudis PV, Grotz MR, Papakostidis C, Dinopoulos H. Operative treatment of displaced fractures of the acetabulum. A meta-analysis. J Bone Joint Surg Br. 2005 Jan;87(1):2-9. PMID 15686228
- [Background] Tannast M, Najibi S, Matta JM. Two to twenty-year survivorship of the hip in 810 patients with operatively treated acetabular fractures. J Bone Joint Surg Am. 2012 Sep 5;94(17):1559-67. doi: 10.2106/JBJS.K.00444. PMID 22992846
- [Background] Clarke-Jenssen J, Roise O, Storeggen SAO, Madsen JE. Long-term survival and risk factors for failure of the native hip joint after operatively treated displaced acetabular fractures. Bone Joint J. 2017 Jun;99-B(6):834-840. doi: 10.1302/0301-620X.99B6.BJJ-2016-1013.R1. PMID 28566406
- [Background] Dodd A, Osterhoff G, Guy P, Lefaivre KA. Assessment of functional outcomes of surgically managed acetabular fractures: a systematic review. Bone Joint J. 2016 May;98-B(5):690-5. doi: 10.1302/0301-620X.98B5.36292. PMID 27143743
- [Background] Ramkumar PN, Haeberle HS, Ramanathan D, Cantrell WA, Navarro SM, Mont MA, Bloomfield M, Patterson BM. Remote Patient Monitoring Using Mobile Health for Total Knee Arthroplasty: Validation of a Wearable and Machine Learning-Based Surveillance Platform. J Arthroplasty. 2019 Oct;34(10):2253-2259. doi: 10.1016/j.arth.2019.05.021. Epub 2019 May 16. PMID 31128890
- [Background] Sanger PC, Hartzler A, Han SM, Armstrong CA, Stewart MR, Lordon RJ, Lober WB, Evans HL. Patient perspectives on post-discharge surgical site infections: towards a patient-centered mobile health solution. PLoS One. 2014 Dec 1;9(12):e114016. doi: 10.1371/journal.pone.0114016. eCollection 2014. PMID 25436912
- [Background] Webb CL, Waugh CL, Grigsby J, Busenbark D, Berdusis K, Sahn DJ, Sable CA; American Society of Echocardiography Telemedicine Collaborators' Group. Impact of telemedicine on hospital transport, length of stay, and medical outcomes in infants with suspected heart disease: a multicenter study. J Am Soc Echocardiogr. 2013 Sep;26(9):1090-8. doi: 10.1016/j.echo.2013.05.018. Epub 2013 Jul 13. PMID 23860093
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Mishra A, Kapoor L, Mishra SK. Post-operative care through tele-follow up visits in patients undergoing thyroidectomy and parathyroidectomy in a resource-constrained environment. J Telemed Telecare. 2009;15(2):73-6. doi: 10.1258/jtt.2008.080808. PMID 19246606
- [Background] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Mobile phone-based telemonitoring for heart failure management: a randomized controlled trial. J Med Internet Res. 2012 Feb 16;14(1):e31. doi: 10.2196/jmir.1909. PMID 22356799
- [Background] Gray RT, Sut MK, Badger SA, Harvey CF. Post-operative telephone review is cost-effective and acceptable to patients. Ulster Med J. 2010 May;79(2):76-9. PMID 21116423